CLINICAL TRIAL: NCT02049528
Title: A Phase 1, Open-Label, Randomized, Crossover Study To Evaluate The Pharmacokinetics Of Single Oral Doses Of Formulated And Non-Formulated CC-122 Capsules And The Effect Of Food On The Pharmacokinetics Of CC-122 In Healthy Adult Male Subjects
Brief Title: Study to Evaluate Pharmacokinetics of Single Oral Doses of Formulated and Non-Formulated CC-122, and Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CC-122-CP-001
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Clinical Pharmacology, Healthy Male Volunteer Study
Keywords: Food Effect; Pharmacokinetic; Healthy; Male
MeSH Terms: interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 mg CC-122 reference capsule formulation (Experimental): 3 mg CC-122 reference capsule given by mouth with 240 mL of room temp tap water
  Interventions: Drug: CC-122
- 3 mg CC-122 test capsule formulation (Experimental): 3 mg CC-122 test capsule give by mouth with 240 mL of room temp tap water
  Interventions: Drug: CC-122
- 3 mg CC-122 test capsule + high fat meal (Experimental): 3 mg CC-122 test capsule given by mouth with 240 mL of room temp tap water approximately 5 minutes after eating a high-fat meal
  Interventions: Drug: CC-122

INTERVENTIONS:
Drug: CC-122 — CC-122
  Arms: 3 mg CC-122 reference capsule formulation
Drug: CC-122 — CC-122
  Arms: 3 mg CC-122 test capsule formulation
Drug: CC-122 — CC-122
  Arms: 3 mg CC-122 test capsule + high fat meal

SUMMARY:
The study is being conducted to compare how long 2 oral formulations (a reference and a test formulation) of CC-122 stays in the body, and whether taking the test formulations with a high-fat meal affects the absorption of that formulation. There will be 3 dosing periods in the study, one for each formulation and one for the test formulation + meal. The subjects will be asked to fast for at least 10 hours before taking the capsule formulations. During one of the periods, the subject will be asked to eat a high-fat meal 30 minutes before being given the capsule to swallow. Subjects will be randomly (by chance) assigned to a treatment sequence which will determine the order in which the subject will receive the reference formulation, the test formulation, and the test formulation + high-fat meal. Blood samples will be taken at intervals during the study to assess the amount of drug at those time points. Blood samples will also be collected at certain time points to determine the levels of special proteins that may help explain how CC-122 work.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy ALL of the following criteria to be enrolled in the study:

  1. Must understand and voluntarily sign a written Informed Consent Document prior to any study-related assessments/procedures being performed and be able to adhere to restrictions and examination schedules.
  2. Must be able to communicate with the Investigator and to understand and adhere to the study visit schedule and other protocol requirements.
  3. Must be a male of any race, aged 18 years of age to 65 years of age (inclusive) at the time of signing the Informed Consent Document.
  4. Has a body mass index (BMI = weight [kilograms (kg)]/(height [m2])) between 18 and 33 kg/m2 (inclusive).
  5. Must be healthy as determined by the Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiograms.

     * Must be afebrile (febrile is defined as body temperature ≥ 38.5 °Celsius or 101.3° Fahrenheit).
     * Systolic blood pressure must be in the range of 90 to 140 millimeters of mercury (mmHg), diastolic blood pressure must be in the range of 50 to 90 mmHg, and pulse rate must be in the range of 45 to 110 beats per minute (bpm).
     * QT interval (Fridericia correction factor) value ≤ 430 milliseconds as measured by an electrocardiogram.
     * Screening and baseline fasting blood glucose must be ≤ 100 milligrams per deciliter (mg/dL) or < 5.6 millimoles per liter (mmol/L), and glycosylated hemoglobin < 6%.
  6. Must practice true abstinence* or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a female of child-bearing potential while participating in this study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.

     * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

       * Must agree to abide by the CC-122 Pregnancy Prevention Risk Management Plan.

Exclusion Criteria:

* The presence of ANY of the following will exclude a subject from enrollment:

  1. History (ie, within 3 years) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders, or known hypersensitivity to a member of the class of immune-mediated inflammatory disease (IMiDs®).
  2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
  3. Use of any prescribed systemic or topical medication within 30 days of the first dose.
  4. Use of any non-prescribed systemic or topical medication (including herbal medicines) within 14 days of the first dose administration (with the exception of vitamin/mineral supplements).
  5. Use of any metabolic enzyme inhibitors or inducers (ie, CYP3A inducers and inhibitors, or St. John's wort) within 30 days of the first dose administration.
  6. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable.
  7. Donated blood or plasma within 8 weeks before the first dose administration.
  8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs).
  9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or positive alcohol screen.
  10. Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg), or hepatitis C antibody, or have a positive result to the test for Human Immunodeficiency Virus antibodies at Screening.
  11. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
  12. Smoke more than 10 cigarettes per day, or the equivalent in other tobacco products (self reported).
  13. Subject has a history of multiple drug allergies (ie, 2 or more).
  14. Subject has any clinical significant allergic disease (excluding non-active hay fever), excluding non-active seasonal allergies and childhood asthma cleared for at least 3 years prior to screening.
  15. Subject received a live vaccine within 90 days of the study drug administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2014-02-02 (Actual); Study Completion 2014-02-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC | up to about 21 days after first dosing
  Area under the plasma concentration-time curve
Pharmacokinetics - Cmax | up to about 21 days after first dosing
  Maximum observed concentration in plasma
Pharmacokinetics - Tmax | up to about 21 days after first dosing
  Time to maximum concentration
Pharmacokinetics - T1/2 | up to about 21 days after first dosing
  Terminal half-life (T1/2)
Pharmacokinetics - CL/F | up to about 21 days after first dosing
  Apparent total body clearance
Pharmacokinetics - Vz/f | up to about 21 days after first dosing
  Apparent volume of distribution

SECONDARY OUTCOMES:
Safety and tolerability | approximately 7-8 weeks
  Safety monitoring will be done by regular adverse event assessment, concomitant medication, clinical laboratory tests, physical exams, ECGs, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene
Locations (1):
- Covance Clinical Development Services, Daytona Beach, Florida, United States